CLINICAL TRIAL: NCT05558644
Title: Characterisation of the Immune Infiltrate and Molecular Features of Thymic Epithelial Tumors Tumors (TETs)
Brief Title: Characterisation of the Immune Infiltrate and Molecular Features of Thymic Epithelial Tumors Tumors (TETs) (IMMUNO-TET)
Acronym: IMMUNO-TET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2022-06
Record Dates: First submitted 2022-09-20; First posted 2022-09-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Cancer
Keywords: thymic epithelial tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm for all patients (Experimental): single arm for all patients tumor samples will be taken for RNA sequencing of epithelial tumour cells during surgery.
  blood samples will be taken for Exome Sequencing (WES) at baseline, during surgery and one month post surgery.
  Interventions: Other: single arm for all patients

INTERVENTIONS:
Other: single arm for all patients — * tumor samples will be taken for RNA sequencing of epithelial tumour cells during surgery.
  * blood samples will be taken for Exome Sequencing (WES) at baseline, during surgery and one month post surgery.

SUMMARY:
The IMMUNO-TET trial aims to assess the feasibility of characterising the immune environment of TETs and the constitutional and somatic molecular profiles of patients with localised thymic epithelial tumour (TET).

DETAILED DESCRIPTION:
In this prospective study, patients undergoing thymectomy and thymomectomy as part of routine care undergo the following care pathway:

1. During the pre-surgical visit (for n = 50 patients): as part of routine care, a blood sample is collected for analysis of CBC, leukocytes, lymphocytes, CRP, ferritinemia, TSH, T3L, T4L, anti-acetycholine receptor antibodies, …CMV, EBV, HSV, HIV serologies, …and HLA class I and class II typing.
2. During thymectomy and thymomectomy surgery, the following samples are taken (for n = 50 patients):

   * 6 blood samples on EDTA tubes are collected at the time of surgery for analyses.
   * 3 fresh samples of the surgical specimen are taken by the pathologist: tumour T, juxta-tumour J and distant D locations for analyses by flow cytometry and RNA sequencing. Anatomopathology blocks/slides are also cut in the same way (tumour T, juxta-tumour J and distant D locations) for additional exploratory analyses.
   * The feasibility of developing patient-derived xenografts (PDX) from TETs will be tested for n = 20 tumor samples. These models will allow to test potential therapeutic agents for this pathology.
3. During the 1st month (+/- 7 days) post-surgery check-up, a blood sample is taken again (for n = 50 patients) for routine care: CBC, leukocytes, lymphocytes, CRP, ferritinemia, anti-acetycholine receptor antibodies and for peripheral immune system analysis at a distance from surgery and for constitutional molecular analysis.

Informed consent is given to participate in this prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with suspicion of localised thymic epithelial tumour.
2. Age ≥ 18 years.
3. Treatment-naïve patient for this disease.
4. Patient with an indication for thymectomy and thymomectomy in one of the partner centers.
5. Signed informed consent form of the patient.

Exclusion Criteria:

1. Neoadjuvant chemotherapy.
2. No social security affiliation.
3. Person under legal protection.
4. Other neoplasia in progress or cured within the last 3 years (except for operated carcinoma in situ).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2026-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Somatic molecular characterisation of TETs | 38 months
  Description of genetic abnormalities in thymic tumours compared to non-tumourous thymic tissue (Whole Exome Sequencing RNA-sequencing technique, DNA Optical mapping);
Characterisation of the immune environment of TETs | 38 months
  Description of immune cells in the tumour environment, description of tumour infiltrating T cells
Establishment of a patient-derived xenograft mouse model. | 38 months
  Patient-derived xenograft mouse model established from thymic tumour.
Molecular characterisation of TETs | 38 months
  Molecular constitutional characterisation of TETs with the technique of the Exome Sequencing (WES) on blood samples of patients with TETs

SECONDARY OUTCOMES:
Genomic characterisation of TETs | 38 months
  WES data analysis constitutional genetic alterations will be performed.
Characterisation of potential alterations in signalling pathways to identify potential therapeutic targets | 38 months
  Molecular analyses will be performed to identify potential alterations in signalling pathways that can be targeted by new therapies.
Identification of potential neoepitopes | 38 months
  Analysis of TETs single-cell RNA-seq data will be performed.
Transcriptomic characterisation of TETs | 38 months
  Transcriptome sequencing analysis will be performed.
Epigenetic characterisation of TETs | 38 months
  Epigenetic characterisation of TETs will be performed by molecular analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Clémence BASSE, MD, Study Director — Institut Curie Paris
Locations (3):
- France (3):
  - Institut Curie Paris, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital FOCH, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).